CLINICAL TRIAL: NCT01193829
Title: Development of Circulating Tumour Cell Molecular Diagnostics Using a Novel Microfluidic Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: PK05/16/10
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Patients With Non-small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Blood will be collected for circulating tumor cells (CTC) using previously optimized methods described by Tan et al. DNA will be extracted from CTC and matching tumor samples (for aim 1) and tested for somatic lung mutations by direct sequencing (2). Germline DNA will be analysed for genes related to putative genetic risks for NSCLC and, for treatment toxicities, for genes related to gefitinib and other chemotherapy metabolic pathways.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC patients

SUMMARY:
1. To compare EGFR mutations between primary non-small cell lung cancer (NSCLC) tumours and corresponding CTCs isolated by a label-free microfluidic device-based system
2. To characterize the association between clinical response in NSCLC patients treated with gefitinib and serial changes in CTC EGFR mutations detected by a label-free microfluidic device-based system

The investigators recently developed a label-free, microfluidic device for capturing circulating tumour cells (CTCs) and acquired a Fluidigm Biomark digital PCR instrument for reliable low-level DNA quantification. The overall aim of this study is to test the feasibility of using these state-of-the-art devices to reliably detect clinically relevant EGFR mutations in CTCs.

DETAILED DESCRIPTION:
For Aim 1, two 5ml pre-treatment blood and corresponding tumor samples will be obtained from NSCLC patients at the National University Health System. Sampling will be organized to avoid the blood samples being the first sample taken after skin puncture to minimize contamination with skin epithelial cells. For the first blood sample, CTCs will be isolated and retrieved using the NUS developed CTC bio-chip according to methods described previously.21 From second blood sample, CTCs will be isolated, fixed on the chip and stained for EpCAM, CD45 and DAPI to assess for cell purity and quantity. DNA will be extracted from the retrieved CTCs and tumour samples, and analyzed exon 19 deletion, L858R and T790M mutations by digital PCR on the Fluidigm Biomark according to methods described previously.23 EGFR mutation status in blood and tumour samples will then be compared for their concordance.

For Aim 2, patients with NSCLC being treated with gefitnib will be approached. Two 5ml blood samples will be obtained pre-treatment (baseline) and then every 4 weeks of treatment (one cycle of gefitinib) from NSCLC patients at the National University Health System.

CTCs will also be obtained and analysed from patients on another protocol receiving gefitinib/ hydroxychloroquine. (B/08/196. A phase II with a lead in phase I study to examine the tolerability, safety profile and efficacy of Hydroxychloroquine and Gefitinib in advanced Non-Small Cell Lung Cancer.) In this study, CTCs are already being collected. Hence the investigators intend to use samples from B/08/196 for CTC analysis using the CTC biochip platform.

For each timepoint, CTCs will be isolated, retrieved and analyzed for EGFR mutation status as described above. Clinical response will be determined using the RECIST criteria.34 Associations between pre-treatment EGFR mutation type quantities and best clinical response will be assessed by Fisher's exact test. Association between trends in EGFR mutation type quantities and tumour size over all treatment cycles will be assessed by observation as performed in the study by Maheswaran et al.9

The investigators plan to analyze 30 patients over one year for both aims of this study. Some cases will have relevant samples (serial blood samples and corresponding tumour) for both aims. The sample size is based on that of the study by Maheshwaran et al.9 and also the likely volume of suitable subjects during 1 year at NUHS. Relevant data for sample size estimation is otherwise lacking. In particular, the frequency of T790M mutations in a relevant patient population is lacking, highlighting the lack of adequate analytical systems for its assessment such as the one proposed in this study.

ELIGIBILITY:
Inclusion Criteria:

* For aim 1:

  * Patients with newly diagnosed non-small cell lung cancer who have not received any systemic therapy such as chemotherapy or targeted therapy.
  * Age 21 years or above
* For aim 2

  * Patients with a diagnosis of non small cell lung cancer
  * Receiving gefitinib as part of their treatment for NSCLC
  * Age 21 years or above

Exclusion Criteria:

* Patients unwilling to provide consent
* Patients, who in the opinion of the investigator, are unable to comply with study requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Tamura K, Okamoto I, Kashii T, Negoro S, Hirashima T, Kudoh S, Ichinose Y, Ebi N, Shibata K, Nishimura T, Katakami N, Sawa T, Shimizu E, Fukuoka J, Satoh T, Fukuoka M; West Japan Thoracic Oncology Group. Multicentre prospective phase II trial of gefitinib for advanced non-small cell lung cancer with epidermal growth factor receptor mutations: results of the West Japan Thoracic Oncology Group trial (WJTOG0403). Br J Cancer. 2008 Mar 11;98(5):907-14. doi: 10.1038/sj.bjc.6604249. Epub 2008 Feb 19. PMID 18283321
- [Background] Sequist LV, Martins RG, Spigel D, Grunberg SM, Spira A, Janne PA, Joshi VA, McCollum D, Evans TL, Muzikansky A, Kuhlmann GL, Han M, Goldberg JS, Settleman J, Iafrate AJ, Engelman JA, Haber DA, Johnson BE, Lynch TJ. First-line gefitinib in patients with advanced non-small-cell lung cancer harboring somatic EGFR mutations. J Clin Oncol. 2008 May 20;26(15):2442-9. doi: 10.1200/JCO.2007.14.8494. Epub 2008 May 5. PMID 18458038